CLINICAL TRIAL: NCT04421677
Title: Safety and Tolerability of Phenylbutyrate in Inclusion Body Myositis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBA in IBM
Record Dates: First submitted 2020-05-18; First posted 2020-06-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-05

CONDITIONS: Inclusion Body Myositis; Sporadic Inclusion Body Myositis
Keywords: Inclusion Body Myositis; IBM; PBA; Phenylbutyrate
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — Phenylbutyrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phenylbutyrate (Experimental): Open-label phenylbutyrate
  Interventions: Drug: Phenylbutyrate Oral Tablet

INTERVENTIONS:
Drug: Phenylbutyrate Oral Tablet — Phenylbutyrate, an orally active chemical chaperone approved by the US Food and Drug Administration for treatment of urea cycle disorders, mimics the function of intracellular molecular chaperones in preventing protein aggregation and oligomerization.
  Other Names: PBA

SUMMARY:
This is a pilot study (phase 1 clinical trial) to evaluate the safety and tolerability of phenylbutyrate in IBM. In this open label study, 10 patients with sporadic inclusion body myositis will be treated with phenylbutyrate (3 gm twice daily) for 3 months. There will be a run-in period, during which certain biomarkers will be measured at baseline and at the end of the run-in period in addition to final measurement at the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill ENMC 2011 diagnostic criteria for IBM
* Age > 18 years
* Women must be post-menopausal (no menses in >12 months) or status post hysterectomy
* Able to give informed consent

Exclusion Criteria:

* Presence of any one of the following medical conditions: chronic infection; chronic renal insufficiency; cancer other than skin cancer less than five years prior; multiple sclerosis or prior episode of central nervous system demyelination; or other chronic serious medical illnesses
* Presence of any of the following on routine blood screening: WBC<3000; Platelets < 100,000; hematocrit < 30%; BUN > 30 mg %; creatine > 1.5 mg%; liver disease with serum albumin < 3 G/DL
* Women who are pregnant or lactating
* History of non-compliance with other therapies
* Coexistence of other muscular disease
* Drug or alcohol abuse within past three months
* Known bleeding disorder
* Known liver disease
* Known congestive heart failure
* Known hypernatremia
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of Phenylbutyrate Measured by Incidence of Adverse Events | Month 3 - Month 6
  Since this is a Phase I pilot trial, the primary outcome will be testing the safety and tolerability of phenylbutyrate in patients with Inclusion Body Myositis. This will be measured by the incidence of adverse events reported in subjects throughout the treatment period of the trial.

SECONDARY OUTCOMES:
Inclusion Body Myositis Functional Rating Scale (IBMFRS) | Month 6
  The IBMFRS is a quickly administered (10-minute) ordinal rating scale (ratings 0-40) used to determine patients' assessment of their capability and independence in 10 functional activities. The higher a subject scores on the scale, the better functional ability the subject has.

CONTACTS AND LOCATIONS:
Overall Officials: Duaa Jabari, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided